CLINICAL TRIAL: NCT04287829
Title: PEMbrolizumab Plus Lenvatinib In Second Line And Third Line Malignant Pleural MEsotheLiomA Patients(PEMMELA)
Brief Title: Pembrolizumab Plus Lenvatinib In Second Line and Third Line Malignant Pleural mesotheLioma Patients
Acronym: PEMMELA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N19PEM
Record Dates: First submitted 2019-11-15; First posted 2020-02-27 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Mesotheliomas Pleural
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pembrolizumab and lenvatinib (Experimental): Patients will receive pembrolizumab 200mg/iv (fixed dose) every 3 weeks and lenvatinib 20mg QD in a three weekly cycle.
  Treatment continues until disease progression by modified RECIST 1.1 for MPM, severe toxicity, serious intercurrent illness, patient request for discontinuation, need or use for any other anti-cancer agent other than protocol treatment, except for palliative radiotherapy, for a maximum period of 35 cycles
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — Infusion
Drug: Lenvatinib — Capsule

SUMMARY:
There is no standard second line treatment in malignant pleural mesothelioma (MPM). Pembrolizumab has shown to be active in in small phase II studies in MPM. Its activity however, is limited, with a response rate up to 20%. Since the arrival of nivolumab plus ipilimumab as first line standard of care treatment in mesothelioma, no treatment options are investigated in this group of patients in the second line. So, there is a need for new treatment combinations with drugs that might exhibit a synergistic interaction with pembrolizumab.

DETAILED DESCRIPTION:
There is no standard second line treatment in malignant pleural mesothelioma (MPM). Pembrolizumab has shown to be active in in small phase II studies in MPM. Its activity however, is limited, with a response rate up to 20%. So, there is a need for new treatment combinations with drugs that might exhibit a synergistic interaction with pembrolizumab. The mechanisms of actions of lenvatinib, which has a broad spectrum of activities, predicts many synergistic interactions with PD-1 blocking. The aim of this study is to characterize the potential clinical activity, toxicity and biomarkers of outcome of pembrolizumab - lenvatinib in patients with recurrent MPM.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed malignant pleural mesothelioma, age at least 18 years
2. Progressive disease after at least 1 and maximal 2 prior systemic treatment lines:

   * Cohort 1: patients, in which one of the lines contains a platinum-based doublet (both cisplatin and carboplatin are allowed) for unresectable MPM (CLOSED)
   * Cohort 2: patients with only in which one of the lines contains nivolumab-ipilimumab immunotherapy as first line treatment for unresectable MPM. No prior chemotherapy.
3. Measurable disease. At least one measurable lesion according to Modified RECIST 1.1 for pleural mesothelioma. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
4. WHO-ECOG performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to date of allocation
5. Adequate organ function
6. Ability to understand the study and give signed informed consent (or legally acceptable representative if applicable) prior to beginning of protocol specific procedures including the approval of the thoracoscopy or transthoracic pleural biopsy before the first treatment cycle and an optional biopsy before the third treatment cycle
7. No presence of clinically relevant treatment-related toxicity from previous chemotherapy, targeted therapy and/or radiotherapy. Note: Participates must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤2 neuropathy may be eligible
8. No active uncontrolled infection, severe cardiac dysfunction (i.e. unstable angina, history of myocardial infarction within the past 12 months prior to screening, congestive heart failure > NYHA II, serious cardiac arrhythmia), unstable peptic ulcer, unstable diabetes mellitus or other seriously disabling condition
9. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mmHg at screening ad no change in hypertensive medication within 1 week before the cycle 1/day1.
10. No prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with another agent agents direct to another stimulatory or co-inhibitory T-cell receptor (eg CTLA-4, OC-40, CD137) or TKI or antibody targeting angiogenesis in the first cohort. Patients who have been treated with autologous tumor cell vaccination (eg. Dendritic cell-based immunotherapy) will be eligible in the first cohort. (First cohort is closed).
11. No concomitant administration to any other experimental drugs under investigation ≤ 4 weeks prior to first admission of pembrolizumab- lenvatinib
12. No prior radiotherapy within 2 weeks before start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids as therapy for radiation induced toxicities. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
13. No major injuries and/or surgery within the past 4 weeks prior to first study dose with incomplete wound healing

Exclusion Criteria:

1. presence of clinically relevant treatment-related toxicity from previous chemotherapy, targeted therapy and/or radiotherapy. Note: Participates must have recovered from all AEs due to previous therapies to 5Grade 1 or baseline. Participants with 52 neuropathy may be eligible
2. active uncontrolled infection, severe cardiac dysfunction (i.e. unstable angina, history of myocardial infarction within the past 12 months prior to screening, congestive heart failure > NYHA II, serious cardiac arrhythmia), unstable peptic ulcer, unstable diabetes mellitus or other seriously disabling condition
3. prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with another agent agents direct to another stimulatory or co-inhibitory T-cell receptor (eg CTLA-4, OC-40, CD137) or TKI or antibody targeting angiogenesis in the first cohort. Patients who have been treated with autologous tumor cell vaccination (eg. Dendritic cell-based imnnunotherapy) will be eligible in the first cohort. (CLOSED)
4. concomitant administration to any other experimental drugs under investigation 5 4 weeks prior to first admission of pembrolizumab- lenvatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate defined by Modified RECIST 1.1 criteria for pleural mesothelioma | Through study completion, an average of 1 year
  Complete response and partial response

SECONDARY OUTCOMES:
Safety of pembrolizumab- lenvatinib | Up to 90 days after last study drug intake
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Describe the disease control rate (DCR) at 3 and 6 months | From date of registration until 6 months
  a percentage of the total number of patients in the study who are evaluable for the primary endpoint who have best overall response of CR or PR or SD.
Objective response rate (ORR) | Assessed up to 60 months
  Number of patients with a partial or complete response
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To describe PFS by independent radiological review

OTHER OUTCOMES:
Immunological status | before study and after 6 weeks of treatment
  The immunological status in the tumors before study and after 6 weeks of treatment with pembrolizumab +lenvatinib. This research will include PD-L1 status, mutational load and other potential biomarkers (e.g. micro vessel density count).

CONTACTS AND LOCATIONS:
Overall Officials: S Burgers, PhD, Principal Investigator — NKI-AvL
Locations (1):
- Antoni van Leeuwenhoekziekenhuis (NKI-AVL), Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Douma LH, van der Noort V, Lalezari F, de Vries JF, Monkhorst K, Smesseim I, Baas P, Schilder B, Vermeulen M, Burgers JA, de Gooijer CJ. Pembrolizumab plus lenvatinib as second-line treatment in patients with pleural mesothelioma (PEMMELA): cohort 2 of a single-arm, phase 2 study. Lancet Oncol. 2025 Dec;26(12):1676-1684. doi: 10.1016/S1470-2045(25)00514-5. PMID 41308680
- [Derived] Douma LH, Lalezari F, van der Noort V, de Vries JF, Monkhorst K, Smesseim I, Baas P, Schilder B, Vermeulen M, Burgers JA, de Gooijer CJ. Pembrolizumab plus lenvatinib in second-line and third-line patients with pleural mesothelioma (PEMMELA): a single-arm phase 2 study. Lancet Oncol. 2023 Nov;24(11):1219-1228. doi: 10.1016/S1470-2045(23)00446-1. Epub 2023 Oct 13. PMID 37844598